CLINICAL TRIAL: NCT03579875
Title: MT2017-17:T Cell Receptor Alpha/Beta T Cell Depleted Hematopoietic Cell Transplantation in Patients With Inherited Bone Marrow Failure (BMF) Disorders
Brief Title: Alpha/Beta TCD HCT in Patients With Inherited BMF Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS161; MT2017-17 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2018-05-25; First posted 2018-07-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Fanconi Anemia; Severe Aplastic Anemia; Myelodysplastic Syndromes; T Cell Receptor Alpha/Beta Depletion; Telomere Biology Disorder; Bone Marrow Failure; Dyskeratosis Congenita; Telomere Biology Disorders
MeSH Terms: conditions — Fanconi Anemia; Anemia, Aplastic; Myelodysplastic Syndromes; Bone Marrow Failure Disorders; Dyskeratosis Congenita | interventions — Whole-Body Irradiation; Cyclophosphamide; fludarabine; Methylprednisolone; Granulocyte Colony-Stimulating Factor; Rituximab; Busulfan; Alemtuzumab; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia (Experimental): Given to:
  * Patients with an unrelated donor or HLA mismatched related donor, regardless of disease type OR
  * Patients with an HLA- identical sibling donor recipient and myelodysplastic features, MDS, or acute leukemia
  Interventions: Drug: Total Body Irradiation (TBI) (Plan 1); Drug: Cyclophosphamide (CY) (Plan 1); Drug: Fludarabine (FLU); Drug: Methylprednisolone (MP); Device: Donor mobilized PBSC infusion; Drug: G-CSF; Drug: Rituximab
- Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia (Experimental): Given to:
  • An HLA-identical sibling donor recipients with single or multi- lineage hematopoietic failure
  Interventions: Drug: Fludarabine (FLU); Drug: Methylprednisolone (MP); Device: Donor mobilized PBSC infusion; Drug: G-CSF; Drug: Cyclophosphamide (CY) (Plan 2); Drug: Rituximab
- Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia (Experimental): Given to:
  * Patients with an unrelated donor or HLA mismatched related donor, regardless of disease type who cannot tolerate TBI
  * Patients with an HLA- identical sibling donor recipient and myelodysplastic features, MDS, or acute leukemia who cannot tolerate TBI
  * Biallelic mutations in FANCD1/BRCA2 who cannot receive TBI
  * Per treating physician preference
  Interventions: Drug: Cyclophosphamide (CY) (Plan 1); Drug: Fludarabine (FLU); Drug: Methylprednisolone (MP); Drug: Rituximab; Drug: Busulfan
- Treatment Plan 4: CY, FLU, and alemtuzumab (Experimental): given to TBD patients with:
  * Bone marrow failure AND
  * Any donor type including haploidentical (4/8) to 8/8-HLA matched related donor, or 7-8/8 HLA-matched unrelated donor Based on historical numbers, it is expected approximately 3 patients would be treated per year. Statistical outcomes will be descriptive.
  Interventions: Drug: Cyclophosphamide (CY) (Plan 1); Drug: Fludarabine (FLU); Drug: Alemtuzumab
- Treatment Plan 5: CY, FLU, melphalan (MEL), and alemtuzumab. (Experimental): given to TBD patients with:
  * Early myelodysplastic features (with or without cytogenetic abnormalities) AND
  * Any donor type including haploidentical (4/8) to 8/8-HLA matched related donor, or 7-8/8 HLA-matched unrelated donor Based on historical numbers, it is expected approximately 2 patients would be treated per year. Statistical outcomes will be descriptive.
  Interventions: Drug: Cyclophosphamide (CY) (Plan 1); Drug: Fludarabine (FLU); Drug: Alemtuzumab; Drug: Melphalan

INTERVENTIONS:
Drug: Total Body Irradiation (TBI) (Plan 1) — 300 cGy with thymic shielding on day -6
  Other Names: TBI
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia
Drug: Cyclophosphamide (CY) (Plan 1) — 10 mg/kg IV daily on days -5, -4, -3, and -2
  Other Names: CY
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia; Treatment Plan 4: CY, FLU, and alemtuzumab; Treatment Plan 5: CY, FLU, melphalan (MEL), and alemtuzumab.
Drug: Fludarabine (FLU) — 35 mg/m2 IV daily on days -5, -4, -3, and -2
  Other Names: FLU
Drug: Methylprednisolone (MP) — 1 mg/kg IV q12h on days -5, -4, -3, -2, and -1
  Other Names: MP
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia
Device: Donor mobilized PBSC infusion — T cell receptor alpha/beta depletion (α/β TCD) peripheral blood stem cell (PBSC) transplantation on day 0
  Other Names: PBSC
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia
Drug: G-CSF — Initiate G-CSF 5mcg/kg per day IV on day +1 (continue until ANC >2.5 x 10^9/L for 3 consecutive days or single day ANC >3000 Arm 1 and Arm 3)
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia
Drug: Cyclophosphamide (CY) (Plan 2) — 5 mg/kg IV daily on days -5, -4, -3, and -2
  Other Names: CY
  Arms: Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia
Drug: Rituximab — 200 mg/m2 IV once on day -1
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia
Drug: Busulfan — Busulfan 0.6 mg/kg if > 4 years old and/or >12 kg (0.8 mg/kg IV if ≤ 4 years old and/or ≤ 12 kg) is given IV over 2 hours every 12 hours for 2 days.
  Other Names: BU
  Arms: Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia
Drug: Alemtuzumab — Alemtuzumab 0.2 mg/kg is given IV over 2 hours daily for 5 days (total dose 1 mg/kg)
  Arms: Treatment Plan 4: CY, FLU, and alemtuzumab; Treatment Plan 5: CY, FLU, melphalan (MEL), and alemtuzumab.
Drug: Melphalan — If available, MEL dosing will be model-based using Bayesian methodology. If Bayesian methodology is unavailable, MEL dosing will be weight-based: MEL 70 mg/m2 for patients ≥10 kg (2.35 mg/kg for patients <10 kg^) IV for one dose over 30 minutes.
  Other Names: MEL
  Arms: Treatment Plan 5: CY, FLU, melphalan (MEL), and alemtuzumab.
Drug: Rituximab — Rituximab will be given once on treatment plans 1-3 on day -1.
  Arms: Treatment Plan 1: TBI 300 , CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 2: CY, FLU, MP, Rituximab in patients with Fanconi Anemia; Treatment Plan 3: BU, Cy, FLU, MP and Rituximab in patients with Fanconi Anemia

SUMMARY:
This is a phase II trial of T cell receptor alpha/beta depletion (α/β TCD) peripheral blood stem cell (PBSC) transplantation in patients with inherited bone marrow failure (BMF) disorders to eliminate the need for routine graft-versus-host disease (GVHD) immune suppression leading to earlier immune recovery and potentially a reduction in the risk of severe infections after transplantation.

ELIGIBILITY:
Patient Selection:

Inclusion Criteria:

For FA patients:

* Diagnosis of Fanconi anemia

  * Age <65 years of age
* Has one of the following risk factors:

  * Severe aplastic anemia (SAA)
  * Myelodysplastic features
  * High risk genotype
  * Immunodeficiency associated with history of recurrent infections
* Karnofsky performance status ≥ 70% if ≥ 16 years of age or Lansky play score ≥ 50% for patients <16 years of age

  * Adequate pulmonary, cardiac and liver function
  * Voluntary written consent (minor assent if appropriate) prior to the performance of any study related procedures not part of standard medical care

For TBD patients:

• Diagnosis of TBD

* Age <70 years of age
* Has one of the following risk factors:
* Severe aplastic anemia (SAA)
* Myelodysplastic features
* Karnofsky performance status ≥ 70% if ≥ 16 years of age or Lansky play score

  ≥ 50% for patients <16 years of age
* Adequate pulmonary, cardiac and liver function
* Voluntary written consent (minor assent if appropriate) prior to the performance of any study related procedures not part of standard medical care

Exclusion Criteria:

* Pregnant or breastfeeding as the treatment used in this study are Pregnancy Category D. Females of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days of study registration
* Active, uncontrolled infection within 1 week prior to starting study therapy
* Malignant solid tumor cancer within previous 2 years

Donor Selection (Inclusion Criteria): meets one of the following match criteria:

* an HLA-A, B, DRB1 matched sibling donor (matched sibling)
* an HLA-A, B, DRB1 matched related donor (other than sibling)
* a related donor mismatched at 1 HLA-A, B, C and DRB1 antigen
* 7-8/8 HLA-A,B,C,DRB1 allele matched unrelated donor per current institutional guidelines Patients and donors are typed for HLA-A and B using serological or molecular techniques and for DRB1 using high resolution molecular typing. If a donor has been selected on the basis of HLA-A, B, C and DRB1 typing as above, preference will be made for donors matched at the HLA-C locus.
* Body weight of at least 40 kilograms and at least 12 years of age
* Willing and able to undergo mobilized peripheral blood apheresis
* In general good health as determined by the medical provider
* Adequate organ function defined as:

  * Hematologic: hemoglobin, WBC, platelet within 10% of upper and lower limit of normal range of test (gender based for hemoglobin)
  * Hepatic: ALT < 2 x upper limit of normal
  * Renal: serum creatinine < 1.8 mg/dl
* Performance of a donor infectious disease screen panel including CMV Antibody, Hepatitis B Surface Antigen, Hepatitis B Core Antibody, Hepatitis C Antibody, HIV 1/2 Antibody, HTLVA 1/2 Antibody, Treponema, and Trypanosoma Cruzi (T. Cruzi) plus HBV, HCV, WNV, HIV by nucleic acid testing (NAT); and screening for evidence of and risks factors for infection with Zika virus, or per current standard institutional donor screen - must be negative for HIV and active hepatitis B
* Not pregnant - females of childbearing potential must have a negative pregnancy test within 7 days of mobilization start
* Voluntary written consent (parent/guardian and minor assent, if < 18 years) prior to the performance of any research related procedure

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
Grade II-IV acute graft versus host disease (GVHD) | Day 100
  incidence of grade II-IV acute graft versus host disease (GVHD)

SECONDARY OUTCOMES:
Neutrophil engraftment | Day 42
  Rate of neutrophil engraftment (defined as the first of three consecutive days after HCT that the patient's absolute neutrophil counts is ≥ 0.5x109 per liter)
Platelet engraftment | Day 42
  Time to platelet engraftment (First of three consecutive days after HCT that the patient's platelet count ≥ 20x10^9 per liter)
Acute graft versus host disease (aGVHD) | Day 100
  Incidence of grade III-IV acute graft versus host disease
Chronic graft versus host disease (cGVHD) | 1 Year after transplant
  Incidence of chronic graft versus host disease after transplant
Regimen related toxicity | 30 Days after transplant
  Incidence of regimen related toxicity based on CTCAE v5
Bacterial, viral and fungal infections | 1 Year after transplant
  Incidence of bacterial, viral and fungal infections
Opportunistic infections | 100 Days after transplant
  Incidence of opportunistic infections
Overall survival (OS) | 1 Year after transplant
  Incidence of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Msc, FRCPC, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States